CLINICAL TRIAL: NCT02806401
Title: Real-time Ultrasound-guided Axillary Venous Catheterization in Pediatric Patients: Comparison With the Landmark Technique Subclavian Vein Catheterization
Brief Title: Ultrasound Guided Axillary Venous Cannulation in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-1603-111-750
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Ultrasound Guided Central Venous Cannulation

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- landmark (Experimental): landmark method_subclavian venous cannulation
  Interventions: Device: landmark
- US_Ax (Active Comparator): ultrasound guided axillary venous cannulation
  Interventions: Device: US_Ax

INTERVENTIONS:
Device: landmark
  Arms: landmark
Device: US_Ax
  Arms: US_Ax

SUMMARY:
The purpose of this prospective randomized study was to compare landmark-subclavian venous access to ultrasound-guided axillary venous access when performed by pediatric anesthesiologists.

DETAILED DESCRIPTION:
Objective: Subclavian vein catheterization may cause various complications. The investigators will compare the real-time ultrasound-guided axillary venous access vs. the landmark method- subclavian venous access in pediatric paticipants. (the needle insertion point of ultrasound-guided axillary venous is axillary vein. and the needle insertion point of landmark method is infraclavicular subclavian vein)

Design: Prospective randomized study.

Setting: Operating room of a tertiary medical center.

Interventions: The investigators will compare the ultrasound-guided axillary vein cannulation (66 paticipants) vs. the landmark method (66 pa- ticipants).

ELIGIBILITY:
Inclusion Criteria:

* surgery under general anesthesia require central venous catheterization

Exclusion Criteria:

* hematoma in central vein central vein anomaly catheterization site infection

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
2nd access success rate | interval between skin penetration and removal of the needle or catheter after central line insertion, an expected average of 120 seconds

SECONDARY OUTCOMES:
1st access success rate | interval between skin penetration and removal of the needle or catheter after central line insertion, an expected average of 120 seconds
3rd access success rate | interval between skin penetration and removal of the needle or catheter after central line insertion, an expected average of 120 seconds
total time | interval between skin penetration and removal of the needle or catheter after central line insertion, an expected average of 120 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea